CLINICAL TRIAL: NCT03283722
Title: Prospective REgistry to Study Clinical OutcomEs of Repair of Mitral ValvEs in South Asia
Brief Title: PRESERVE-MITRAL Post-Market Registry
Status: Completed | Type: Observational
Sponsor: Medtronic Cardiac Surgery (Industry)
Responsible Party: Sponsor
Other Study IDs: MDT16016SUR002
Record Dates: First submitted 2017-08-09; First posted 2017-09-14 (Actual); Results first posted 2025-02-11 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Mitral Valve Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Profile 3D™ and CG Future® annuloplasty system — Patients suffering from mitral valve disease and indicated for a mitral valve repair procedure with Profile 3D™ and CG Future® annuloplasty system as part of standard of care, in accordance with the product label indications (instructions for use), contraindications, and warnings

SUMMARY:
The objective of this registry is to gather data on the clinical outcomes of Medtronic mitral repair products (Profile 3D™ and CG Future® annuloplasty systems) in the approved intended use up to 12 months from the day of procedure

DETAILED DESCRIPTION:
There is limited local evidence on mitral repair products in South Asia and a prospective post market registry will provide real world data on clinical outcomes.

Patients suffering from mitral valve disease and indicated for a mitral valve repair procedure with Profile 3D™ and CG Future® annuloplasty system as part of standard of care, in accordance with the product label indications (instructions for use), contraindications, and warnings will be considered for study participation.

PRESERVE-Mitral Registry is a prospective non-randomized, non-interventional, post-market registry

The objective of this registry is to gather data on the clinical outcomes of Medtronic mitral repair products (Profile 3D™ and CG Future® annuloplasty systems) in the approved intended use up to 12 months from the day of procedure

This clinical trial information was submitted voluntarily under the applicable law and, therefore, certain submission deadlines may not apply. (That is, clinical trial information for this applicable clinical trail was submitted under section 402(j)(4)(A) of the Public Health Service Act and 42CFR 11.60 and is not subject to the deadlines established by sections 402(j)(2) and (3) of the Public Heath Service Act or 42 CRF 11.24 and 11.44.)

ELIGIBILITY:
Inclusion Criteria:

1. Patients with valvular insufficiency and/or stenosis and indicated for the reconstruction and/or remodeling of pathological mitral valves with Profile 3D™ and CG Future® annuloplasty systems
2. Indications and contraindications provided in the product Instructions for Use
3. Subject is 18 years of age or older
4. The patient or his/her Legally Authorized Representative (LAR) has been informed about the nature of the registry and the patient informed consent for study participation has been obtained prior to performing any study-related procedures from the subject or Legally Authorized Representative, as per applicable local requirements

Exclusion Criteria:

1. Contraindications as per instructions-for-use (IFU):

   1. Heavily calcified valves
   2. Valvular retraction with severely reduced mobility
   3. Active bacterial endocarditis
2. Aortic valve replacement as concomitant procedure
3. Already participating in another clinical study, possibly leading to bias and jeopardizing the scientific appropriate assessment of the study endpoints

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suffering from mitral valve disease and indicated for a mitral valve repair procedure with Profile 3D™ and CG Future® annuloplasty system as part of standard of care, in accordance with the product label indications (instructions for use), contraindications, and warnings
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2017-04-10 (Actual); Primary Completion 2021-02-10 (Actual); Study Completion 2021-02-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vinay Rajan, Ph.D, Study Chair — Medtronic
Locations (12):
- National Heart Foundation Hospital & Research Institute, Dhaka, Bangladesh
- India (10):
  - U. N. Mehta Institute of Cardiology and Research Centre, Ahmedabad, Gujarat
  - SAL Hospital & Medical Institute, Ahmedabad, Gujarat
  - EPIC Hospital, Ahmedabad, Gujarat
  - Sri Jayadeva Institute of Cardiovascular Sciences & Research, Bangalore, Karnataka
  - Narayana Institute of Cardiac Sciences, Bangalore, Karnataka
  - Amrita Institute of Medical Sciences and Research Center, Kochi, Kerala
  - P.D. Hinduja National Hospital and Medical Research Centre, Mumbai, Maharashtra
  - The Madras Medical Mission, Chennai, Tamil Nadu
  - G. Kuppuswamy Memorial Hospital, Coimbatore, Tamil Nadu
  - CARE Hospitals, Hyderabad, Telangana
- Manmohan Cardiothoracic Vascular and Transplant Center, Kathmandu, Nepal

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Mitral Valve Repair With Profile 3D™ or CG Future® Annuloplasty System: Subjects requiring mitral valve repair and are intended to receive either Profile 3D™ or CG Future® annuloplasty device.
Period: Overall Study
Arm/Group | Mitral Valve Repair With Profile 3D™ or CG Future® Annuloplasty System
Started | 200
Completed | 180 (Completed definition included those subjects were successfully implanted and followed.)
Not Completed | 20

BASELINE CHARACTERISTICS:
Population: 200 total subjects enrolled, 184 had an attempted; and, 180 were successfully implanted and followed. Data reported is for the Successfully Implanted (IMP) cohort n=180.
Arm/Group | Mitral Valve Repair With Profile 3D™ or CG Future® Annuloplasty System
Number analyzed (Participants) | 180
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Data reported is for the Successfully Implanted (IMP) cohort n=180.
  years | 50.4 (15.0)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Data reported is for the Successfully Implanted (IMP) cohort n=180.
  Participants
    Female | 65
    Male | 115
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants] — Population: Data reported is for the Successfully Implanted (IMP) cohort n=180.
  participants
    Bangladesh | 23
    Nepal | 13
    India | 144
Weight [Mean (Standard Deviation); unit: kg] — Demographics and baseline characteristics are summarized for the Enrolled and Successfully Implanted analysis sets including subject weight. Population: Data reported is for the Successfully Implanted (IMP) cohort n=180.
  kg | 61.4 (12.2)
Height [Mean (Standard Deviation); unit: cm] — Demographics and baseline characteristics including height are summarized for the Enrolled and Successfully Implanted analysis sets Population: Data reported is for the Successfully Implanted (IMP) cohort n=180.
  cm | 161.4 (9.5)
NYHA Classification [Count of Participants; unit: Participants] — The New York Heart Association (NYHA) Functional Classification is a system for defining cardiac disease and related functional limitations into four broad categorizations:
  NYHA Classification:
  Class I: Subjects with cardiac disease but without resulting limitations of physical activity.
  Class I: Subjects with cardiac disease resulting in slight limitation of physical activity.
  Class III: Subjects with cardiac disease resulting in marked limitation of physical activity.
  Class IV: Subjects with cardiac disease resulting in inability to carry on any physical activity without discomfort. Population: Data reported is for the Successfully Implanted (IMP) cohort n=180, there are 8 subjects that did not have a reported NYHA classification.
  Participants
    No Heart Failure: number analyzed (Participants) | 172
    No Heart Failure | 0
    Class I: number analyzed (Participants) | 172
    Class I | 6
    Class II: number analyzed (Participants) | 172
    Class II | 91
    Class III: number analyzed (Participants) | 172
    Class III | 66
    Class IV: number analyzed (Participants) | 172
    Class IV | 9
Cardiac Rhythm [Count of Participants; unit: Participants] — Population: Data reported is for the Successfully Implanted (IMP) cohort n=180. Two subjects did not have an ECG reported at baseline.
  Participants
    Atrial Fibrillation: number analyzed (Participants) | 178
    Atrial Fibrillation | 10
    Atrial Flutter: number analyzed (Participants) | 178
    Atrial Flutter | 2
    Normal Sinus Rhythm: number analyzed (Participants) | 178
    Normal Sinus Rhythm | 154
    Other: number analyzed (Participants) | 178
    Other | 12
Surgical History [Count of Participants; unit: Participants] — Population: Data reported is for the Successfully Implanted (IMP) cohort n=180.
  Participants
    Coronary artery bypass graft (CABG) | 1
    Percutaneous transluminal coronary angioplasty (PTCA) | 5
    Other | 9
Risk Factors [Count of Participants; unit: Participants] — Population: Data reported is for the Successfully Implanted (IMP) cohort n=180.
  Participants
    Atrial Fibrillation | 1
    Congestive Heart Failure | 21
    Coronary Artery Disease | 87
    Diabetes Mellitus | 60
    Pulmonary Hypertension | 9
    Renal Insufficiency, Dialysis | 2
    Systemic Hypertension | 54
    Other | 34
Mitral Valve Pathophysiology [Count of Participants; unit: Participants] — Population: Data reported is for the Successfully Implanted (IMP) cohort n=180.
  Participants
    Barlow's Disease | 7
    Congenital Pathophysiology | 2
    Ischemic Pathophysiology | 76
    Marfan's Syndrome | 1
    Rheumatic Pathophysiology | 72
    Myxomatous | 23
Mitral Valve Regurgitation [Count of Participants; unit: Participants] — Population: Data reported is for the Successfully Implanted (IMP) cohort n=180.
  Participants
    Moderate | 29
    Moderate to Severe | 14
    Severe | 137

OUTCOME MEASURES:

1. Primary Outcome: Improvement in Mitral Regurgitation (MR) Grade at 12-months Post Procedure
Description: This is determined by assessing the level of mitral valve regurgitation using echo, in subjects at 12-months post-procedure compared to the level at baseline. The levels of regurgitation, level 0-4, correspond to the American Society of Echocardiography (ASE) guidelines ranging from no MR, Mild MR, Moderate MR, Moderate- to-Severe MR and Severe MR. A percentage number is calculated to reflect how many participants had an MR improvement.
Time Frame: 12 months
Population: Data reported is for the Successfully Implanted (IMP) cohort n=180.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Mitral Valve Repair With Profile 3D™ or CG Future® Annuloplasty System
Number analyzed (Participants) | 180
percentage of participants | 97.8 [93.8 to 99.6]

2. Primary Outcome: All Cause Mortality
Description: All deaths occurring from any cause 12-months post procedure
Time Frame: 12 months
Measure: Number; unit: participants
Arm/Group | Mitral Valve Repair With Profile 3D™ or CG Future® Annuloplasty System
Number analyzed (Participants) | 180
participants | 6

3. Secondary Outcome: Percentage of Participants With Improvement in MR Grade at Discharge and First Follow-up (3-6 Months)
Description: This was determined by assessing the level of mitral valve regurgitation using hemodynamic performance, in subjects at discharge and 3-6 months post-procedure compared to the level at baseline. The levels of regurgitation, level 0-4, correspond to the ASE guidelines ranging from no MR, Mild MR, Moderate MR, Moderate-to-Severe MR and Severe MR
Time Frame: At discharge from hospital (up to 7 days) and at first follow-up (3-6month)
Population: Of the 180 implanted subjects, 161 returned for the first follow-up visit at 3-6 months and had an echo performed, primarily due to standard of care practices at participating facilities.
Measure: Number (95% Confidence Interval); unit: percentage of patients with improved MR
Arm/Group | Mitral Valve Repair With Profile 3D™ or CG Future® Annuloplasty System
Number analyzed (Participants) | 180
percentage of patients with improved MR
  Discharge | 100 [98.0 to 100]
  3-6 month: number analyzed (Participants) | 161
  3-6 month | 97.5 [93.8 to 99.3]

4. Secondary Outcome: Improvement in NYHA Functional Class at Discharge, First Follow-up (3-6 Months) and Second Follow-up (12-months) Compared to Baseline.
Description: The percentage of subjects with an improved New York Heart Association NYHA functional class using a two-sided 95% exact binomial confidence internal measured at discharge, 3-6 months, and 12-months post-procedure and compared to baseline.
Time Frame: At discharge from hospital (up to 7 days), at first follow-up (3-6months), and at the second follow-up (12 months)
Population: Subject follow-up based on standard of care at participating centers
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Mitral Valve Repair With Profile 3D™ or CG Future® Annuloplasty System
Number analyzed (Participants) | 180
percentage of participants
  Discharge: number analyzed (Participants) | 169
  Discharge | 73.4 [66.0 to 79.9]
  3-6 Months: number analyzed (Participants) | 155
  3-6 Months | 84.5 [77.8 to 89.8]
  12 Months | 83.8 [76.7 to 89.5]

5. Secondary Outcome: Hospitalization for Heart Failure at 6 Months and at 12 Months Post Procedure
Description: Subjects who have a non-elective hospital admission for signs and symptoms related to heart failure that results in a one night stay (i.e., where the admission date and the discharge date differ by at least one calendar day)
Time Frame: 6 months and 12 months post procedure
Population: Data reported is for the Successfully Implanted (IMP) cohort n=180. Data was not reported for 19 subjects at the 6 month visit and 70 subjects at the 12 month visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Mitral Valve Repair With Profile 3D™ or CG Future® Annuloplasty System
Number analyzed (Participants) | 180
Participants
  6 Months: number analyzed (Participants) | 161
  6 Months | 4
  12 Months: number analyzed (Participants) | 110
  12 Months | 1

6. Secondary Outcome: Mitral Valve Re-intervention at Discharge, 6 Months and at 12 Months Post Procedure
Description: Subject leaving the operating theater with an implanted Profile 3DTM or CG Future® annuloplasty system and later undergo any surgical or percutaneous interventional catheter procedure that repairs, otherwise alters or adjusts, or replaces the previously implanted annuloplasty system is considered a reoperation
Time Frame: At discharge from hospital (up to 7 days), at first follow-up (3-6months), and at the second follow-up (12 months)
Population: Data reported is for the Successfully Implanted (IMP) cohort n=180.
Measure: Count of Participants; unit: Participants
Arm/Group | Mitral Valve Repair With Profile 3D™ or CG Future® Annuloplasty System
Number analyzed (Participants) | 180
Participants
  Discharge | 0
  Discharge through 6 months | 0
  12 months | 0

7. Secondary Outcome: Stroke at 6 Months and at 12 Months Post Procedure
Description: Subjects had an acute episode of focal or global neurological dysfunction caused by brain, spinal cord, or retinal vascular injury as a result of hemorrhage or infarction, where the neurological dysfunction lasts for greater than 24-hours
Time Frame: 6 months and 12 months post procedure
Population: Data reported is for the Successfully Implanted (IMP) cohort n=180. Data was not reported for 17 subjects at 6 months and 68 subjects at 12 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Mitral Valve Repair With Profile 3D™ or CG Future® Annuloplasty System
Number analyzed (Participants) | 180
Participants
  6 month: number analyzed (Participants) | 163
  6 month | 2
  12 month: number analyzed (Participants) | 112
  12 month | 0

8. Secondary Outcome: New Onset of Atrial Fibrillation, as Evaluated Through Follow up ECG at Discharge, First Follow up (3-6months) and at Second Follow up (12 Months)
Description: New onset of AF is defined as when the subject did not present with prior history of AF at baseline nor was AF detected at baseline visit, but AF did manifest post procedure and was either diagnosed during the study visits (discharge, 3-6 months or 12 months visit) or was otherwise diagnosed during the duration of subject participation in the study. The incidence of new onset AF will be evaluated at discharge, first follow up (3-6 months) and at second follow up (12 months). This endpoint is analyzed for the Successfully Implanted (IMP) cohort and provided as a Kaplan-Meier analysis.
Time Frame: At discharge from hospital, (up to 7 days), at first follow-up (3-6month), and at the second follow-up (12 months)
Population: Data reported is for the Successfully Implanted (IMP)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Mitral Valve Repair With Profile 3D™ or CG Future® Annuloplasty System
Number analyzed (Participants) | 169
percentage of participants
  Discharge: number analyzed (Participants) | 161
  Discharge | 3.6 [1.6 to 7.8]
  3-6 Months: number analyzed (Participants) | 149
  3-6 Months | 4.8 [2.4 to 9.6]
  12 months: number analyzed (Participants) | 107
  12 months | 4.8 [2.1 to 10.8]

9. Secondary Outcome: Number of Attempts Required for Procedural Success
Description: Number of surgical attempts required for procedural implant success
Time Frame: Procedure (defined as the date of the first attempted procedure through subject leaving the operating theater with an implanted Profile 3D or CG Future annuloplasty system)
Population: Data reported is for the Successfully Implanted (IMP) cohort n=180.
Measure: Count of Participants; unit: Participants
Groups:
- Mitral Valve Repair With Profile 3D™ or CG Future® Annuloplasty System: Number of attempts required for procedural success, and bypass time as a measure of procedural complexity
Arm/Group | Mitral Valve Repair With Profile 3D™ or CG Future® Annuloplasty System
Number analyzed (Participants) | 180
Participants
  One Attempt | 177
  Two Attempts | 3

10. Secondary Outcome: Total Bypass Time During the Implant Procedure
Description: Total time a subject is on bypass time as a measure of procedural complexity
Time Frame: During the procedure as measured by standard operating procedures at the sites
Population: Data reported is for the Successfully Implanted (IMP) cohort n=180.
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Mitral Valve Repair With Profile 3D™ or CG Future® Annuloplasty System
Number analyzed (Participants) | 180
Minutes | 125.1 (47.0)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Mitral Valve Repair With Profile 3D™ or CG Future® Annuloplasty System
All-Cause Mortality (participants affected / at risk) | 6/180
Serious Adverse Events (participants affected / at risk) | 24/180
Other Adverse Events (participants affected / at risk) | 0/180
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mitral Valve Repair With Profile 3D™ or CG Future® Annuloplasty System (N=180)
Arrhythmia (Cardiac disorders) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 1 (1)
Atrial Flutter (Cardiac disorders) | 1 (1)
Cardiac Arrest (Cardiac disorders) | 1 (1)
Cardiac Failure (Cardiac disorders) | 2 (2)
Cardiac Failure Congestive (Cardiac disorders) | 3 (6)
Cardiopulmonary Failure (Cardiac disorders) | 1 (1)
Left Ventricular Dysfunction (Cardiac disorders) | 1 (1)
Right Ventricular Dysfunction (Cardiac disorders) | 1 (1)
Death (General disorders) | 2 (2) — Unknown cause
Pyelonephritis (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1)
Cerebrovascular Accident (Nervous system disorders) | 2 (2)
Acute Kidney Injury (Renal and urinary disorders) | 1 (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Decubitus Ulcer (Skin and subcutaneous tissue disorders) | 1 (1)
Renal Transplant (Surgical and medical procedures) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-04-10): https://cdn.clinicaltrials.gov/large-docs/22/NCT03283722/Prot_SAP_000.pdf